CLINICAL TRIAL: NCT00940771
Title: Equivalence of Boosted Atazanavir Based Regimens and Currently Effective HAART Regimens With Other PI's/NNRTI's in HIV+ Children and Adolescents With Elevated Lipid Levels
Brief Title: Equivalence of Boosted Atazanavir Based Regimens and Currently Effective HAART Regimens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Phoenix Children's Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Janice Piatt, Medical Director, Bill Holt Clinic, Phoenix Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCH 09-004
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Results first posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Pediatric HIV; HIV Infections
Keywords: HIV; Lipids; Atazanavir; Pediatric; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- boosted Atazanavir (Experimental): Boosted Atazanavir was switched for the PI or NNRTI in the patients regimen
  Interventions: Drug: Boosted Atazanavir

INTERVENTIONS:
Drug: Boosted Atazanavir — Boosted Atazanavir, once a day dose adjusted for child's weight for 6 months.
  Other Names: Reyataz

SUMMARY:
The hypothesis for this study is whether a treatment regimen containing Atazanavir in combination with Ritonavir will work as well as other regimens containing a protease inhibitor and/or a Non-nucleoside Reverse Transcriptase Inhibitor (NNRTI) at controlling HIV disease in children who are HIV+ and have high cholesterol or high triglycerides. . In this study, children who have high cholesterol or high triglycerides as a result of their HIV medicines, will have the PI or NNRTI in their medication regimen changed to Atazanavir, which is a PI in combination with a low dose of Ritonavir (another PI). Atazanavir has been shown in adults to result in lower cholesterol and triglycerides than other PI's and NNRTI's. The dose of Atazanavir and Ritonavir will be according to the Package Insert for this drug that is FDA approved for children. They will continue taking the other medications from the pre-study regimen. Children will take study drug for 24 weeks, and will be able to continue study drug after the study using commercially available drug. Lab tests and a physical exam will be undertaken at 4 weeks, 12 weeks and 24 weeks after starting study drug to determine how effective the new drug is and to monitor for possible side effects.

DETAILED DESCRIPTION:
The primary objective of this study is to determine if Atazanavir and Ritonavir together will be as effective as the child's previous regimen in keeping the level of virus in the blood stream at such a low level it can't be found and whether that combination will be as effective as the previous regimen in keeping the infection fighting cells in the blood at the same level.

Secondary objectives will be:

* To determine if cholesterol and triglyceride levels drop in children switching to Atazanavir and Ritonavir from other medication regimens.
* To evaluate if Atazanavir and Ritonavir result in an increase in patient satisfaction and patient reported adherence and a decrease in symptoms related to medication side effects.

Inclusion Criteria are:

* On the same medication regimen at least 3 months
* Weight equal to or greater than 25kg
* Able to swallow pills or willing to learn
* Have a parent or guardian willing and able to sign informed consent
* Not be taking a medication which interacts with Atazanavir
* Not be currently taking Sustiva

ELIGIBILITY:
Inclusion Criteria:

* HIV positive children with elevated lipid levels
* on stable HAART for at least 3 months (defined to be on the same regimen with viral load < 1000 for 6 months prior to baseline visit).
* Weight equal to or greater than 25kg
* Able to swallow pills or willing to learn

Exclusion Criteria:

* Patients with underlying hepatitis B or C viral infections
* Previously demonstrated clinically significant hypersensitivity (eg, Stevens-Johnson syndrome, erythema multiforme, or toxic skin eruptions) to any of the components of Reyataz® (atazanavir).
* Taking other medications that are highly dependent on CYP3A or UGT1A1 for clearance

  * Ergot medicines: dihydroergotamine, ergonovine, ergotamine, and methylergonovine such as Cafergot®, Migranal®, D.H.E. 45®, ergotrate maleate, Methergine®, and others (used for migraine headaches).
  * Orap® (pimozide, used for Tourette's disorder).
  * Propulsid® (cisapride, used for certain stomach problems).
  * Triazolam, also known as Halcion® (used for insomnia).
  * Midazolam, also known as Versed® (used for sedation), when taken by mouth.
  * Camptosar® (irinotecan, used for cancer).
  * Crixivan® (indinavir, used for HIV infection).
  * Cholesterol-lowering medicines Mevacor® (lovastatin) or Zocor® (simvastatin).
  * Rifampin (also known as Rimactane®, Rifadin®, Rifater®, or Rifamate®).
  * St. John's wort (Hypericum perforatum), an herbal product sold as a dietary supplement,
  * Viramune® (nevirapine, used for HIV infection).
  * Vfend® (voriconazole).
* Patients with grade 3 or higher elevations in transaminases (> 10 X ULN)
* Women of Childbearing Potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period.
* Women who are pregnant or breastfeeding.
* Women with a positive pregnancy test.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2009-08-26 (Actual); Primary Completion 2013-10-16 (Actual); Study Completion 2016-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Piatt, MD, Principal Investigator — Phoenix Children's Hospital
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric patients with elevated cholesterol were recruited from a Pediatric HIV Clinic between April 8, 2009 and May 1, 2013.
Period: Pre-Entry
Arm/Group | Boosted Atazanavir
Started | 10
Completed | 10
Not Completed | 0
Period: 4 Weeks
Arm/Group | Boosted Atazanavir
Started | 10
Completed | 10
Not Completed | 0
Period: 12 Weeks
Arm/Group | Boosted Atazanavir
Started | 10
Completed | 10
Not Completed | 0
Period: 24 Weeks
Arm/Group | Boosted Atazanavir
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Boosted Atazanavir
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 9.5 [6 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
CD4 [Mean (Standard Deviation); unit: cells/uL] | 1233.1 (473.8)
Viral Load [Mean (Standard Deviation); unit: copies/ml] | 2.3 (7.3)
Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 214.3 (31.6)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 288.5 (253.9)

OUTCOME MEASURES:

1. Primary Outcome: Non-fasting Cholesterol
Time Frame: 4 Weeks, 12 weeks, 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Boosted Atazanavir
Number analyzed (Participants) | 10
mg/dL
  Week 4 | 187.2 (30.0)
  Week 12 | 178.5 (38.1)
  Week 24 | 181.5 (29.3)
Statistical Analysis 1: Comparison: Boosted Atazanavir; Test type: Other — Friedman's Test; p = .006, Friedman's Test; 3 degrees of freedom; Chi Square = 12.3
Statistical Analysis 2: Comparison: Boosted Atazanavir; Nul lHypothesis that there is no difference between specific time points; Test type: Other — Post Hoc testing Post hoc Wilcoxon Signed Rank tests; p = .007, Wilcoxon Signed Rank; Z=-2.701

2. Primary Outcome: Non-fasting Triglycerides
Time Frame: 4 weeks, 12 weeks, 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Boosted Atazanavir
Number analyzed (Participants) | 10
mg/dL
  Week 4 | 240.5 (107.2)
  Week 12 | 195.5 (93.8)
  Week 24 | 193.3 (106.5)
Statistical Analysis 1: Comparison: Boosted Atazanavir; Test type: Other — Friedman's test with 3 df; p = .356, Friedman's Test; 3 degrees of freedom

3. Secondary Outcome: Viral Load
Description: Number of participants with undetectable viral load
Time Frame: 4 weeks, 12 weeks, 24 weeks
Population: Number of patients with undetectable viral load
Measure: Count of Participants; unit: Participants
Arm/Group | Boosted Atazanavir
Number analyzed (Participants) | 10
Participants
  Week 4 | 10
  Week 12 | 9
  Week 24 | 9
Statistical Analysis 1: Comparison: Boosted Atazanavir; The null hypothesis was that there was a difference. We were looking for no difference between before and after switch; Test type: Other; p = .801, Friedman's test; 3 degrees of freedom; Chi-square = 1.0 — 1.0 is the actual calculated Chi-X value, not the p value

4. Secondary Outcome: CD4 Count
Time Frame: 4 Weeks, 12 weeks, 24 weeks
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Boosted Atazanavir
Number analyzed (Participants) | 10
cells/uL
  Week 4 | 1214.3 (476.8)
  Week 12 | 1151.9 (442.7)
  Week 24 | 1120.0 (413.2)
Statistical Analysis 1: Comparison: Boosted Atazanavir; Test type: Other — Friedman's test; p = .075, Friedman's test — a priori threshold for statistical significance 0.05; 3 degrees of freedom

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events V 1.0, December 2004, Clarification August 2009 was used to grade labs and symptoms that were reported at week 4, week 12 and week 24 visits.
Arm/Group | Boosted Atazanavir
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boosted Atazanavir (N=10)
Pansinusitis (Infections and infestations) | 1 (1) — Pansinusitis requiring hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boosted Atazanavir (N=10)
Pain, neck and face (Blood and lymphatic system disorders) | 1 (1) — Pain grade 2 associated with parotitis
Fever (General disorders) | 2 (2) — Fever grade 2 associated with Parotitis or Upper Respiratory Infection
Pain, throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) — pain grade 2 associated with Upper Respiratory Infection
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Cough grade 2 associated with Upper Respiratory Infection
Vomiting (Gastrointestinal disorders) | 1 (1) — Grade 3 vomiting associated with parotitis
Laboratory Abnormality (Gastrointestinal disorders) | 1 (3) — Elevated Bilirubin, grade 3

LIMITATIONS AND CAVEATS:
Small sample size Non fasting lipid levels Large variety of prior treatment regimens

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No